CLINICAL TRIAL: NCT04484818
Title: A Phase III Double Blinded Study of Early Intervention After RADICAl ProstaTEctomy With Androgen Deprivation Therapy With or Without Darolutamide vs. Placebo in Men at Highest Risk of Prostate Cancer Metastasis by Genomic Stratification (ERADICATE)
Brief Title: Testing the Addition of Darolutamide to Hormonal Therapy (Androgen Deprivation Therapy [ADT]) After Surgery for Men With High-Risk Prostate Cancer, The ERADICATE Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA8183; NCI-2020-02383 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8183 (Other: ECOG-ACRIN Cancer Research Group); EA8183 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Goserelin; Leuprolide; luprolide acetate gel depot; Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (ADT, placebo) (Active Comparator): Patients receive goserelin acetate, leuprolide acetate, or triptorelin via injection every 3 months for 12 months (4 injections), every 4 months for 12 months (3 injections), or every month for 12 months (12 injections) in the absence of disease progression or unacceptable toxicity. Patients also receive a placebo four times daily (QID) for 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Drug: Triptorelin
- Arm B (ADT, darolutamide) (Experimental): Patients receive goserelin acetate, leuprolide acetate, or triptorelin via injection every 3 months for 12 months (4 injections), every 4 months for 12 months (3 injections), or every month for 12 months (12 injections) in the absence of disease progression or unacceptable toxicity. Patients also receive darolutamide QID for 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Darolutamide; Drug: Goserelin Acetate; Drug: Leuprolide Acetate; Other: Quality-of-Life Assessment; Drug: Triptorelin

INTERVENTIONS:
Drug: Darolutamide — Given PO
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; ODM 201; ODM-201
  Arms: Arm B (ADT, darolutamide)
Drug: Goserelin Acetate — Given via injection
  Other Names: ZDX; Zoladex
Drug: Leuprolide Acetate — Given IV
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Drug: Placebo Administration — Given PO
  Arms: Arm A (ADT, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Triptorelin — Given via injection
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY-25650; CL-118,532; Detryptoreline

SUMMARY:
This phase III trial compares the effect of adding darolutamide to ADT versus ADT alone after surgery for the treatment of high-risk prostate cancer. ADT reduces testosterone levels in the blood. Testosterone is a hormone made mainly in the testes and is needed to develop and maintain male sex characteristics, such as facial hair, deep voice, and muscle growth. It also plays role in prostate cancer development. Darolutamide blocks the actions of the androgens (e.g. testosterone) in the tumor cells and in the body. Giving darolutamide with ADT may work better in eliminating or reducing the size of the cancer and/or prevent it from returning compared to ADT alone in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether 12 months of androgen deprivation therapy (ADT) and darolutamide improves metastasis-free survival (MFS) compared to 12 months of ADT plus placebo in men with high risk prostate cancer (defined by Cancer of the Prostate Risk Assessment Post-surgical [CAPRA-S] score >= 3 and a high Decipher score (>= 0.6) [C3+D+]) who have undergone radical prostatectomy.

SECONDARY OBJECTIVES:

I. To determine whether 12 months of ADT and darolutamide improves recurrence-free survival (RFS) compared to 12 months of ADT plus placebo in men with high-risk prostate cancer that have undergone radical prostatectomy.

II. To determine whether 12 months of ADT and darolutamide improves event-free survival (EFS) compared to 12 months of ADT plus placebo in men with high-risk prostate cancer that have undergone radical prostatectomy.

III. To determine whether 12 months of ADT and darolutamide improves overall survival (OS) compared to 12 months of ADT plus placebo in men with high-risk prostate cancer that have undergone radical prostatectomy.

IV. To determine the rate of testosterone recovery and time to testosterone recovery in each treatment arm.

V. To evaluate the safety and tolerability of ADT and darolutamide.

CORRELATIVE OBJECTIVES FOR EXPLORATORY BIOMARKERS:

I. To discover a novel gene expression signature in the Decipher transcriptome platforms that is predictive of clinical outcome, as defined by the primary and secondary objectives of this study, in response to ADT by intensification with darolutamide versus ADT alone.

II. To assess the prevalence of subclasses of established transcriptome expression signatures and prospectively validate their predictive value for ADT response, these include: (i) androgen (AR) activity (ii) Basal-luminal subtyping based on modified PAM50, and (iii) ADT score.

III. To assess whether the spectrum of high Decipher scores (0.6-1.0), prostate-specific antigen (PSA) levels at presentation and post-radical prostatectomy (RP) and final pathology variables affect the response and outcome to ADT and darolutamide.

QUALITY OF LIFE (QOL) OBJECTIVES:

I. To compare overall quality of life, measured by Functional Assessment of Cancer Therapy-Prostate (FACT-P) total score, at 18 months between the two arms. (Primary) II. To compare the change in overall quality of life, measured by FACT-P total score, from baseline to 18 months between the two arms. (Secondary) III. To compare patient-reported fatigue (Functional Assessment of Chronic Illness Therapy [FACIT]-Fatigue scores) at 12 months between the two treatment arms. (Secondary) IV. To compare the change in subjective patient-reported cognitive function (FACT-Cognitive [Cog]) from baseline to 12 months between the treatment arms. (Exploratory) V. To compare subjective patient-reported cognitive function (FACT-Cog scores) at 12 months between the two treatment arms. (Exploratory)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive goserelin acetate, leuprolide acetate, or triptorelin via injection every 3 months for 12 months (4 injections), every 4 months for 12 months (3 injections), or every month for 12 months (12 injections) in the absence of disease progression or unacceptable toxicity. Patients also receive a placebo four times daily (QID) for 52 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive goserelin acetate, leuprolide acetate, or triptorelin via injection every 3 months for 12 months (4 injections), every 4 months for 12 months (3 injections), or every month for 12 months (12 injections) in the absence of disease progression or unacceptable toxicity. Patients also receive darolutamide QID for 52 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION (STEP 0)
* Patient must have undergone a radical prostatectomy (RP) and must be registered to step 0 of this study at least 6 weeks after but not more than 16 weeks after their radical prostatectomy
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0- 2
* Patient with a prior or concurrent malignancy within 5 years of registration, whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* For patients with no previous Decipher score: Tumor tissue specimen from prostatectomy must be available and ready to be shipped
* INCLUSION CRITERIA FOR RANDOMIZATION (STEP 1)
* For patients who have previously had Decipher score performed by Decipher Biosciences, they must have score of >= 0.6
* For patients who did not have a Decipher score previously performed by Decipher Biosciences, they must have had a Decipher score of >= 0.6 assessed from the prostatectomy specimen submitted
* For patients who did not have a Decipher score previously performed by Decipher Biosciences, patients must also have a CAPRA-S score >= 3. The CAPRA-S score is calculated by assigning points for PSA in ng/mL, surgical margin status, seminal vesicle invasion, and extra-capsular extension. Lymph node involvement will serve as an exclusion criteria and will not count towards CAPRA-S inclusion score. A CAPRA-S score is not required for patients who had a Decipher score previously performed by Decipher Biosciences
* Patient must have an undetectable PSA (< 0.2ng/mL) obtained within 2 weeks prior to randomization
* Leukocytes >= 3,000/mcL (obtained within 4 weeks prior to registration)
* Absolute neutrophil count >= 1,000/mcL (obtained within 4 weeks prior to registration)
* Platelets >= 75,000/mcL (obtained within 4 weeks prior to registration)
* Total bilirubin =< institutional upper limit of normal (ULN) (obtained within 4 weeks prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (obtained within 4 weeks prior to registration)
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 (obtained within 4 weeks prior to registration)

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION (STEP 0)
* Patient must not have any previous treatment with androgen deprivation therapy (ADT), chemotherapy, or other physician prescribed systemic therapy for treatment of their prostate cancer
* Patient must not have pathologic evidence of pelvic lymph node involvement
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association class III and IV heart failure), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* EXCLUSION CRITERIA FOR RANDOMIZATION (STEP 1)
* Patient must not have pre or post-operative radiographic evidence of cancer recurrence or metastasis by abdominal and pelvic imaging (computed tomography [CT] abdomen/pelvis, whole body magnetic resonance imaging [MRI], MRI abdomen/pelvis, or equivalent, AND bone scan) which must be done before or after prostatectomy prior to randomization. If pre-operative risk does not indicate a need for bone scan, post-operative Decipher score of >= 0.6 indicates increased risk of metastatic disease and may be used to obtain CT abdomen/pelvis and bone scan prior to randomization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival (MFS) | From randomization to development of metastatic disease or death, whichever occurs first, assessed up to 36 months
  The primary comparison will be an intention-to-treat analysis of all randomized patients. The method of Kaplan and Meier will be used to characterize the time-to-event endpoints, and a logrank test will be used to compare these endpoints across treatments.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | From randomization to any of the MFS events, pelvic lymph node recurrence or detectable prostate-specific antigen (PSA) (PSA >= 0.2 ng/mL, confirmed by a second PSA of the same level or higher), whichever occurs first, assessed up to 36 months
  The method of Kaplan and Meier will be used to characterize the time-to-event endpoints, and a logrank test will be used to compare these endpoints across treatments.
Event-free survival | From randomization to any of the RFS events, treatment with salvage radiation therapy with or without systemic therapy, or initiation of systemic therapy for presumed recurrence, whichever occurs first, assessed up to 36 months
  The method of Kaplan and Meier will be used to characterize the time-to-event endpoints, and a logrank test will be used to compare these endpoints across treatments.
Overall survival | From randomization to death by any cause or date last known alive, assessed up to 36 months
  The method of Kaplan and Meier will be used to characterize the time-to-event endpoints, and a logrank test will be used to compare these endpoints across treatments.
Testosterone recovery rate | At time of disease progression, assessed up to 36 months
  Exact binomial confidence intervals will be used to describe the proportions of patients with testosterone recovery in each arm.
Time to testosterone recovery | From randomization to a return of serum testosterone level to greater than or equal to lower limit of normal for the testosterone assay, assessed up to 36 months
  The method of Kaplan and Meier will be used to characterize the time-to-event endpoints, and a logrank test will be used to compare these endpoints across treatments.
Incidence of adverse events | Up to 78 weeks
  Toxicity will be defined using the Common Terminology Criteria for Adverse Events version 5.0.
Change in quality of life: Functional Assessment of Cancer Therapy (FACT) | Baseline up to 18 months
  Will be assessed by the Functional Assessment of Cancer Therapy (FACT) - Prostate, FACT - Cognitive, and Functional Assessment of Chronic Illness Therapy - Fatigue. Fatigue instruments at baseline, 6, 12 and 18 months, and descriptive statistics will be used to characterize quality of life over time in each arm. Each item is answered on a 5-point Likert-type scale, where a value of 0 indicates the statement is not applicable, and a value of 5 indicates the statement is applicable to the respondent. Subgroup analysis will be performed among patients who receive adjuvant radiation therapy and patients who do not receive adjuvant radiation therapy in each arm. Mixed effect models will be constructed as an exploratory analysis to estimate the time profile of quality of life assessments in the two arms and to evaluate treatment-by-time interactions.
Overall quality of life: Functional Assessment of Cancer Therapy (FACT) | At 18 months
  Will be assessed by the Functional Assessment of Cancer Therapy (FACT) - Prostate total score. The total score can range from 0 to 156, where a higher value indicates a better quality of life. Mixed effect models will be constructed as an exploratory analysis to estimate the time profile of quality of life assessments in the two arms and to evaluate treatment-by-time interactions.
Change in Functional Assessment of Cancer Therapy (FACT) - Prostate score | Baseline up to 18 months
  A paired t test will be used to compare Functional Assessment of Cancer Therapy (FACT) - Prostate scores at these two time points in each arm. The total score can range from 0 to 156, where a higher value indicates a better quality of life. A two-sample t test will be performed to compare the changes in FACT - Prostate scores from baseline to 18 months between the two arms. Mixed effect models will be constructed as an exploratory analysis to estimate the time profile of quality of life assessments in the two arms and to evaluate treatment-by-time interactions.

OTHER OUTCOMES:
Cognitive function | At 12 months (completion of treatment)
  Will be measured between the two arms by Functional Assessment of Cancer Therapy (FACT) - Cognitive. The FACT-Cognitive has four subscales: perceived cognitive impairments (PCI), perceived cognitive abilities, impact of perceived cognitive impairment on quality of life, and comments from others on cognitive function. Summary statistics will be used to describe each subscale at each time point and the PCI subscale score, which ranges from 0-72, where higher values indicate better quality of life, at 12 months will be the primary measurement of this analysis. Bonferroni correction will be employed for the 3 follow-up time points of interest (6, 12, and 18 months) to make the analysis conservative. Mixed effect models will be constructed as an exploratory analysis to estimate the time profile of quality of lifeassessments in the two arms and to evaluate treatment-by-time interactions.
Change in cognitive function | Baseline up to 12 months (completion of treatment)
  Will be measured between the two arms by Functional Assessment of Cancer Therapy (FACT) - Cognitive. The FACT-Cognitive has four subscales: perceived cognitive impairments (PCI), perceived cognitive abilities, impact of perceived cognitive impairment on quality of life, and comments from others on cognitive function. Summary statistics will be used to describe each subscale at each time point and the PCI subscale score, which ranges from 0-72, where higher values indicate better quality of life, at 12 months will be the primary measurement of this analysis. Bonferroni correction will be employed for the 3 follow-up time points of interest (6, 12, and 18 months) to make the analysis conservative. Mixed effect models will be constructed as an exploratory analysis to estimate the time profile of quality of life assessments in the two arms and to evaluate treatment-by-time interactions.
Identification of novel gene expression signatures | Up to 36 months
  The associations between the gene expression signatures and clinical outcomes will be assessed by Cox proportional hazards models and logrank test.
Prognostic value of established signatures | Up to 36 months
  Will include androgen receptor activity, basal-luminal subtyping by modified PAM50 and androgen deprivation therapy score using Cox proportional hazards models. Similar analysis will be performed to evaluate the prognostic value of luminal-basal subtype. The treatment-by-subtype interaction will also be assessed. For androgen deprivation therapy score, patients will be categorized into either low or high androgen deprivation therapy score using a cutoff of 0.36.
Decipher scores | Up to 36 months
  Will be associated with MFS as well as disease characteristics. Cox proportional hazards models will be performed with adjustment for important disease characteristics, including prostate-specific antigen, Gleason score, disease stage, pathology of the radical prostatectomy specimen, etc. Decipher score could be categorized into a few risk groups and the Akaike information criterion method will be used to determine the optimal number of cutoff points. To assess whether treatment effect is affected by Decipher score levels, the treatment-by-Decipher interactions will be included in the model as well. Decipher scores range from 0.00 to 1.00, where higher values indicate higher risk disease.
Genome-wide alterations | Up to 36 months
  Prostate cancer specimens will be banked for future studies to perform genome-wide alterations in coding and non-coding deoxyribonucleic acid sequences. To identify the genetic alterations that are associated with development of metastasis, Cox proportional hazards models and logrank test will be used. The analysis will focus on actionable alterations first. The treatment-by-alteration interactions will also be assessed to determine whether response to darolutamide is affected by distinct genomic subgroups. Ultimately the findings on gene expression signatures and deoxyribonucleic acid alterations will be assessed in the models simultaneously to identify subsets of patients who might benefit most from the treatment of ADT with or without darolutamide.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia K Morgans, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (115):
- United States (115):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - Hartford Hospital, Hartford, Connecticut
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - GenesisCare USA - Clarkston, Clarkston, Michigan
  - GenesisCare USA - Farmington Hills, Farmington Hills, Michigan
  - GenesisCare USA - Macomb, Macomb, Michigan
  - GenesisCare USA - Madison Heights, Madison Heights, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin